CLINICAL TRIAL: NCT05809492
Title: Use of A-STEP Test in Cystic Fibrosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MAR.FTR.AD2
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: patients between the ages of 18-50 with a diagnosis of cystic fibrosis FEV1 >70%, FEV1 40-70% and FEV1 <40% who are clinically stable are patients with cystic fibrosis Deciency FEV1 >70%, FEV1 <40%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with a diagnosis of cystic fibrosis, FEV1(functional expiratory volume)< 40% (Experimental): calculation of the maximum exercise capacity using the a-step test
  Interventions: Other: step test
- Patients with a diagnosis of cystic fibrosis, FEV1(functional expiratory volume)< 40-70% (Experimental): calculation of the maximum exercise capacity using the a-step test
  Interventions: Other: step test
- Patients with a diagnosis of cystic fibrosis, FEV1(functional expiratory volume)> 70% (Experimental): calculation of the maximum exercise capacity using the a-step test
  Interventions: Other: step test

INTERVENTIONS:
Other: step test — The step speed of 18 steps/min was chosen for the first level because it is suitable for all subjects and prevents them from being too fast at the end of the test.
  the slow standardized initial tempo at Level 1 of 72 beats/min allowed familiarity with the coordinated cascading technology of the tests (step up and down in time with the metronome beat). Regular replacement of the leading leg was encouraged to prevent unilateral leg fatigue and November muscle pain.
  pwCF selected 1-minute stage times for each level in accordance with the maximum exercise test (CPET) recommendations in 18; at each new level, the test speed was increased by two steps / minute to ensure a progressive change in exercise parameters; a suitable end test time of 16 minutes was achieved along with an initial speed of 18 steps/min. The fast pace of 194 beats/min (48 steps/min at Level 16), which was eventually reached, it was physically possible to perform safely.

SUMMARY:
The exercise test provides prognostic information about clinical outcomes and quality of life to optimize care for cystic fibrosis patients (pwCF). The exercise test identifies the causes of exercise restriction, adverse exercise reactions, and exercise-related symptoms. The results help to determine and evaluate the impact of exercise programs at PWCF. Peak oxygen uptake (VO2peak) is a prognostic measure of maximum exercise capacity that usually worsens as CF lung disease progresses.

The recommended gold standard exercise test at PWCF is a cardiopulmonary exercise test (CPET) performed on a loop ergometer to assess VO2peak and cardiopulmonary responses to exercise. the recommended incremental protocol, consisting of 1-minute phases, should reach VO2peak within 8-12 minutes. Trained operators perform cpets with complex and expensive laboratory equipment, and it is inaccessible and little used by many people internationally.

Step tests are low-cost, portable, easily standardized and require minimal space to perform. The 3-Minute Step Test (3MST) is an externally paced test for the assessment of exercise tolerance set at 30 steps/minute for 3 minutes. In adults with CF, 3MST is useful for assessing oxygen desaturation and predicting future increased use of healthcare services. Limitations include the ceiling effect in less severe CF lung disease, and it is very difficult for some with more advanced lung disease.

An incremental maximum A-STEP step test has been developed to assess exercise capacity in the CF lung disease December, without floor or ceiling effects, within clinical space constraints and the need for strict infection prevention.

A-STEP is a new incremental maximum step test to assess exercise capacity in PWCF without floor or ceiling effects, as an alternative field test to CPET.

DETAILED DESCRIPTION:
The exercise test provides prognostic information about clinical outcomes and quality of life to optimize care for cystic fibrosis patients (pwCF). The exercise test identifies the causes of exercise restriction, adverse exercise reactions, and exercise-related symptoms. The results help to determine and evaluate the impact of exercise programs at PWCF. Peak oxygen uptake (VO2peak) is a prognostic measure of maximum exercise capacity that usually worsens as CF lung disease progresses.

The recommended gold standard exercise test at PWCF is a cardiopulmonary exercise test (CPET) performed on a loop ergometer to assess VO2peak and cardiopulmonary responses to exercise. the recommended incremental protocol, consisting of 1-minute phases, should reach VO2peak within 8-12 minutes. Trained operators perform cpets with complex and expensive laboratory equipment, and it is inaccessible and little used by many people internationally.

Step tests are low-cost, portable, easily standardized and require minimal space to perform. The 3-Minute Step Test (3MST) is an externally paced test for the assessment of exercise tolerance set at 30 steps/minute for 3 minutes. In adults with CF, 3MST is useful for assessing oxygen desaturation and predicting future increased use of healthcare services. Limitations include the ceiling effect in less severe CF lung disease, and it is very difficult for some with more advanced lung disease.

An incremental maximum A-STEP step test has been developed to assess exercise capacity in the CF lung disease December, without floor or ceiling effects, within clinical space constraints and the need for strict infection prevention.

A-STEP is a new incremental maximum step test to assess exercise capacity in PWCF without floor or ceiling effects, as an alternative field test to CPET.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with cystic fibrosis between the ages of 18 and 50 Dec
* FEV 1 value must be at least 20%
* Being clinically stable (no hospitalization for at least 30 days, no history of acute exacerbations, no changes in maintenance therapy)

Exclusion Criteria:

* Having evidence of febrile illness
* Hemoptysis
* Uncontrolled asthma
* Pneumothorax
* Cardiac, vascular and renal comorbidities
* Pulmonary hypertension
* CF-related diabetes
* Body mass index <18 kg/m2
* Pregnancy
* Inability to follow instructions safely

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Calculation of the maximum exercise capacity using the step test in cystic fibrosis patients | 18 minute
  Calculation of the maximum exercise capacity using the step test in cystic fibrosis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Mamara Üniversitesi Tıp Fakültesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No